CLINICAL TRIAL: NCT03181165
Title: Impact of a Pharmacist-led Therapeutic Nutritional Intervention on Medications and Glucose Control in Type 2 Diabetes
Brief Title: Pharmacist-led Therapeutic Nutritional Intervention in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mitacs (Industry); Pharmasave (Unknown)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-01539
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Diet Modification
Keywords: Low-carbohydrate; Low calorie; Energy restricted

STUDY DESIGN:
Intervention Model Description: Pragmatic effectiveness trial of diet intervention led by community pharmacists versus treatment-as-usual waitlist control.
Masking Description: Participants will know group assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-carbohydrate Therapeutic Nutrition (Experimental): A 12-week low-carbohydrate, energy-restricted diet will be administered using a combination of pre-packaged foods and whole foods from pre-specified lists.
  Interventions: Behavioral: Low-carbohydrate Therapeutic Nutrition
- Treatment-as-usual waitlist control (No Intervention): Participants will receive standard lifestyle advice to follow a low-fat, low-sugar, high fibre diet and aim to accumulate 150 minutes of moderate activity per week.

INTERVENTIONS:
Behavioral: Low-carbohydrate Therapeutic Nutrition — The pharmacist or pharmacy lifestyle coach will work with the participant to develop a diet plan that is low in carbohydrate and energy-restricted based on personal preferences and characteristics. A combination of pre-packaged low-carbohydrate foods and whole foods from pre-specified lists will be used.
  Arms: Low-carbohydrate Therapeutic Nutrition

SUMMARY:
Type 2 diabetes represents a significant burden to both the individual and our healthcare system. Individuals with type 2 diabetes are typically prescribed one or more glucose-lowering medications, many of which have undesirable side effects (e.g., nausea, risk of cardiovascular complications, weight gain) and cost our healthcare system a lot of money. An alternative strategy to lower blood glucose is to consume a low-carbohydrate diet. However, adjusting medications after choosing to follow a low-carbohydrate diet can be difficult. Delivering a low-carbohydrate diet through pharmacists could circumvent this difficulty in medications adjustment because pharmacists are trained to adjust medications. In this study the investigators will determine whether type 2 diabetes patients can reduce medications and improve blood glucose by following a low-carbohydrate, low-calorie diet under the direction of a pharmacist.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 30 and 75, have type 2 diabetes mellitus diagnosed by a physician, are taking one or more glucose-lowering medications, have a BMI ≥30, have no contraindications to following low-carbohydrate, energy-restricted, high-protein diet, and can read and speak English.

Exclusion Criteria:

Exlcusion criteria are:

1. Recent (within the last 2 years) diagnosis of coronary heart disease, stroke, or a heart attack.
2. Unstable cardiovascular disorder.
3. History of liver disease.
4. History of kidney disease or impaired renal function.
5. Previously undergone bariatric surgery.
6. Multiple sclerosis or other diagnosed neurological disease.
7. Currently pregnant or lactating, or planning on becoming pregnant in the next 12 months.
8. Any form of cancer within the last 5 years.
9. Body mass index (BMI) of <30.
10. Dietary restrictions that do not allow you to follow a low-carbohydrate, energy-restricted, high-protein diet (e.g., vegan, food allergies).
11. Any sensitivities to the ingredients in the pre-packaged foods

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants not on glucose-lowering medications | 12 weeks
  Number of individuals taking no medications divided by the total number of participants.

SECONDARY OUTCOMES:
Hemoglobin A1C | 12 weeks
  Blood test to measure glucose control
Reduction in glucose-lowering medications | 12 weeks
  Reduction in total dose of glucose-lowering medications
Body mass index | 12 weeks
  Body mass in kilograms divided by height in meters squared.
Waist circumference | 12 weeks
  Waist circumference in centimeters
Body fat percentage | 12 weeks
  Body fat percentage measured by bioelectrical impedance analysis
Body mass | 12 weeks
  Body mass in kg
Health related quality of life | 12 weeks
  Short-form (SF)-20 questionnaire
Reduction in non-glucose lowering medications | 12 weeks
  Dose of medications other than glucose-lowering
Blood lipid profile | 12 weeks
  triglycerides, HDL and LDL cholesterol
Fasting insulin | 12 weeks
  Fasting insulin
Fasting C-peptide | 12 weeks
  fasting C-peptide
C-reactive protein | 12 weeks
  Fasting high-sensitivity C-reactive protein
Liver enzymes | 12 weeks
  liver alanine amino transferase, aspartate aminotransferase, gamma-gluatmyl transpeptidase
Fasting plasma glucose | 12 weeks
  Fasting plasma glucose
Systolic Blood Pressure | 12 weeks
  Systolic Blood Pressure measured by automatic cuff
Diastolic Blood Pressure | 12 weeks
  Diastolic Blood Pressure measured by automatic cuff

OTHER OUTCOMES:
Habitual physical activity | 12 weeks
  Godin leisure-time exercise questionnaire
Energy intake | Baseline, 6 weeks, and 12 weeks
  3-day diet record
Macronutrient intake | Baseline, 6 weeks, and 12 weeks
  3-day diet record
Intervention Satisfaction | 12 weeks
  Satisfaction with intervention delivery questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Little, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual values will be reported in figures if applicable.

REFERENCES:
- [Derived] Durrer C, Islam H, Cen HH, Garzon MDM, Lyu X, McKelvey S, Singer J, Batterham AM, Long JZ, Johnson JD, Little JP. A secondary analysis of indices of hepatic and beta cell function following 12 weeks of carbohydrate and energy restriction vs. free-living control in adults with type 2 diabetes. Nutr Metab (Lond). 2024 May 27;21(1):29. doi: 10.1186/s12986-024-00807-x. PMID 38797835
- [Derived] Durrer C, McKelvey S, Singer J, Batterham AM, Johnson JD, Gudmundson K, Wortman J, Little JP. A randomized controlled trial of pharmacist-led therapeutic carbohydrate and energy restriction in type 2 diabetes. Nat Commun. 2021 Sep 10;12(1):5367. doi: 10.1038/s41467-021-25667-4. PMID 34508090
- [Derived] Durrer C, McKelvey S, Singer J, Batterham AM, Johnson JD, Wortman J, Little JP. Pharmacist-led therapeutic carbohydrate restriction as a treatment strategy for type 2 diabetes: the Pharm-TCR randomized controlled trial protocol. Trials. 2019 Dec 27;20(1):781. doi: 10.1186/s13063-019-3873-7. PMID 31881991